CLINICAL TRIAL: NCT04843098
Title: Phase I/II Study of the PI3K Inhibitor TL117 Alone and in Combination With Paclitaxel in Patients With Relapsed/Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of TL117 in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Junde Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TL-117-202001
Record Dates: First submitted 2021-03-19; First posted 2021-04-13 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm, open label (Experimental): Phase 1a: All subjects receiving TL117 alone (20-120 mg); Phase 1b: All subjects receiving TL117 (MTD-1 or MTD) plus Paclitaxel; Phase 2: All subjects receiving TL117 in combination with Paclitaxel at RP2D
  Interventions: Drug: TL117; Drug: Paclitaxel

INTERVENTIONS:
Drug: TL117 — TL117 capsules orally once daily
Drug: Paclitaxel — Paclitaxel (80 mg/m2) administered intravenously (IV) on Days 1, 8, and 15 of a 28-day treatment cycle.

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetic and efficacy of TL117 plus paclitaxel in patients with recurrent or metastatic head and neck cancer.

DETAILED DESCRIPTION:
This is a Phase 1/2 open label, single arm study, and is divided into three phases: the single-agent dose-escalation phase Ia trial, the TL117 plus paclitaxel dose-escalation phase Ib trial, and the open label, multicenter phase 2 trial of TL117 plus paclitaxel.

Adverse events and dose limiting toxicities will be assessed from the first dose of study drug though day 28. When the maximum tolerated dose (MTD) of TL117 plus paclitaxel is determined, additional patients will be treated at the defined RP2D dose until occurrence of unacceptable toxicity, disease progression or withdrawal of consent or death.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old for Phase 1a, 18-75 years old for Phase 1b and 2;
2. Histologically and/or cytologically confirmation of recurrent/metastatic squamous cell carcinoma of the head and neck;
3. At least one evaluable or measurable tumor lesion;
4. Adequate performance status;
5. A minimum life expectancy of > 3 months;
6. Adequate cardiac, kidney, and liver function;
7. Willingness of all subjects of childbearing potential to use acceptable methods of birth control;

Exclusion Criteria:

1. Any chemotherapy, radiotherapy, targeted therapy, immunotherapy, endocrine therapy and other systematic anti-tumor therapies within 4 weeks prior to the first dose of the study drug (some exceptions apply)
2. Prior or current PI3K inhibitor therapy;
3. Type 1 or type 2 diabetes requiring antihyperglycemic medication;
4. Major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the first dose, or required elective surgery during the study period;
5. Any unresolved toxicities from prior therapy greater than Grade 1;
6. Inability to swallow, or serious gastrointestinal absorption conditions;
7. History of immunodeficiency;
8. Active central nervous system metastases;
9. Active hepatitis B or C virus infection;
10. Uncontrolled active infection;
11. Serious cardiovascular disease；
12. Clinically uncontrollable effusion in the third space;
13. Known allergy and/or contraindications to paclitaxel;
14. Known alcohol or drug dependence;
15. Mental disorders or poor compliance;
16. Pregnant or lactating women;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Phase Ia -Dose Limiting Toxicity (DLT) of TL117 treatment | From time of the first dosing to time of Cycle 1 Day 28（each cycle is 28 days）
  Per DLT criteria as defined in protocol
Phase Ib -Dose Limiting Toxicity (DLT) of TL117 plus paclitaxel combination treatment | From time of the first dosing to time of Cycle 1 Day 28（each cycle is 28 days）
  Per DLT criteria as defined in protocol
Phase II - Objective response rate (ORR) | Every 8 weeks from date of first treatment until date of last treatment up to 12 months
  Objective response rate (ORR): percentage of patients with best overall response of complete response (CR) and partial response (PR) according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No